CLINICAL TRIAL: NCT00000741
Title: A Controlled Randomized Trial to Study the Efficacy of Adjunctive Methylprednisolone for the Treatment of Pneumocystis Carinii Pneumonia (PCP) in Pediatric AIDS Patients
Brief Title: The Safety and Effectiveness of Methylprednisolone in the Treatment of Pneumocystis Carinii Pneumonia (PCP) in Children With AIDS
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Upjohn (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: ACTG 170
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: Pneumonia, Pneumocystis carinii; Acquired Immunodeficiency Syndrome; Methylprednisolone
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Methylprednisolone

INTERVENTIONS:
Drug: Methylprednisolone

SUMMARY:
To determine the effect of methylprednisolone on respiratory failure in HIV-infected patients with presumed or confirmed pneumocystis carinii pneumonia who are stratified for presence or absence of respiratory failure at the time of randomization to the study.

DETAILED DESCRIPTION:
HIV-infected children are randomized to receive adjunctive therapy with intravenous methylprednisolone or placebo. Treatment is administered for 10 days. Primary antipneumocystis therapy with TMP/SMX or systemic pentamidine is selected by the individual investigator and given for 21 days. Patients are stratified at the time of randomization by the presence or absence of respiratory failure.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Recombinant erythropoietin and any FDA-approved cytokine for management of anemia.
* Antiretroviral agents.

Patients must have:

* Documented HIV infection.
* PCP.
* No more than 36 hours of prior primary therapy for confirmed or presumed PCP.

Prior Medication:

Allowed:

* Up to 35 hours of primary therapy for confirmed or presumed PCP.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Demonstrated intolerance to steroids.
* Requirement for steroids at greater than physiological doses for other medical conditions.

Ages: 28 Days to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dankner WM, Study Chair; Bozzette S, Study Chair; Spector SA, Study Chair
Locations (6):
- United States (6):
  - UCSD Med Ctr / Pediatrics / Clinical Sciences, La Jolla, California
  - Chicago Children's Memorial Hosp, Chicago, Illinois
  - St Louis Univ School of Medicine, St Louis, Missouri
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Duke Univ Med Ctr, Durham, North Carolina

REFERENCES:
- [Background] National Institutes of Health-University of California Expert Panel for Corticosteroids as Adjunctive Therapy for Pneumocystis Pneumonia. Consensus statement on the use of corticosteroids as adjunctive therapy for pneumocystis pneumonia in the acquired immunodeficiency syndrome. N Engl J Med. 1990 Nov 22;323(21):1500-4. doi: 10.1056/NEJM199011223232131. No abstract available. PMID 2136587